CLINICAL TRIAL: NCT00354159
Title: Reducing Decompensation Events Utilizing Intracardiac Pressures in Patients With Chronic HF (REDUCEhf)
Brief Title: Reducing Decompensation Events Utilizing Intracardiac Pressures in Patients With Chronic Heart Failure (HF) (REDUCEhf)
Acronym: REDUCEhf
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 103
Record Dates: First submitted 2006-07-19; First posted 2006-07-20 (Estimated); Results first posted 2012-08-09 (Estimated); Last update posted 2012-08-09 (Estimated); Status verified 2012-08

CONDITIONS: Heart Failure
Keywords: Implantable cardioverter defibrillator; Intracardiac pressures
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment Arm (Experimental): Physicians have access to device-based hemodynamic monitor information to guide patient management
  Interventions: Device: Implantable Hemodynamic Monitor (Chronicle® IHM), and IHM in combination with single chamber ICD (Chronicle ICD)
- Control Arm (Placebo Comparator): Physicians do not have access to device-based hemodynamic monitor information to guide patient management
  Interventions: Device: Implantable Hemodynamic Monitor (Chronicle® IHM), and IHM in combination with single chamber ICD (Chronicle ICD)

INTERVENTIONS:
Device: Implantable Hemodynamic Monitor (Chronicle® IHM), and IHM in combination with single chamber ICD (Chronicle ICD) — Surgical implantation of hemodynamic device (IHM), or IHM/ICD, and intracardiac leads.
  Other Names: Chronicle® IHM, Chronicle® ICD

SUMMARY:
The purpose of this clinical research study is to evaluate the safety and effectiveness of the investigational implantable hemodynamic monitor (IHM), and of the IHM in combination with an implantable cardioverter defibrillator (ICD). The investigational IHM has the ability to record and report the force with which the heart pumps blood (heart pressures). When combined with the ICD, the device has the additional ability to send a strong electrical impulse, or shock, to the heart when it detects dangerously fast heartbeats to return it to a normal rhythm. The IHM and IHM/ICD are implanted surgically just under the skin in the upper chest area. This study will also determine how doctors use the information related to heart pressures in the management of heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with heart failure that only sometimes interferes with daily activities (New York Heart Association [NYHA] Class II (1)) or subjects with heart failure which severely limits daily activities (NYHA Class III (2)) at baseline
* Subject has appropriate medical therapy for heart failure (such as diuretic, angiotensin-converting enzyme (ACE) inhibitor or angiotensin receptor blocker (ARB) and beta blocker) for at least three months prior to the baseline evaluation.
* Subject has been on stable medications maximized to the subject's tolerance of ACE or ARB and beta blockers as determined by the study investigator for at least 30 days prior to baseline evaluation. (Stable is defined as no more than a 100% increase or a 50% decrease in dose.) If a subject is intolerant of ACE, ARB or beta blockers documented evidence must be available.
* Subject has had at least one heart failure-related hospitalization or at least one heart failure-related emergency department or urgent care visit necessitating heart failure-related intravenous therapy (e.g. diuretic administration) within 12 months prior to the baseline evaluation
* To be considered for Chronicle ICD: Subject has, or is at risk of having, a heart beat that is too fast and his/her doctor has determined he/she needs an implantable cardioverter defibrillator (ICD).

  1. Class II Subjects with cardiac disease resulting in slight limitation of physical activity. They are comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea, or angina.
  2. Class III Subjects with cardiac disease resulting in marked limitation of physical activity. They are comfortable at rest. Less than ordinary activity causes fatigue, palpitation, dyspnea, or angina.

Exclusion Criteria:

* Subjects with severe heart failure who should always be resting (NYHA Class IV(3)) or Stage D(4) refractory heart failure.
* Subjects with severe renal dysfunction.
* Subjects with severe non-cardiac condition limiting 12-month survival.
* Subjects in concurrent studies that may confound the results.

  (3)Class IV Subjects with cardiac disease resulting in inability to carry on any physical activity without discomfort. Symptoms of heart failure or the anginal syndrome may be present even at rest. If any physical activity is undertaken, discomfort is increased.

  (4)Stage D refractory heart failure: Patients who have marked symptoms at rest despite maximal medical therapy (e.g., those who are recurrently hospitalized or cannot be safely discharged from the hospital without specialized interventions)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 442 (Actual)
Dates: Start 2006-04; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phillip Adamson, MD, Study Chair — Oklahoma Heart Hospital; Michael Gold, MD, Study Chair — Medical University of South Carolina
Locations (52):
- United States (52):
  - University of Alabama at Birmingham (UAB), Birmingham, Alabama
  - Scripps Green Hospital, La Jolla, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Long Beach Memorial, Long Beach, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Doctors Medical Center Modesto, Modesto, California
  - Yale University, School of Medicine, New Haven, Connecticut
  - Christiana Care Hospital, Newark, Delaware
  - University of FL Shands, Gainesville, Florida
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Crawford Long/Emory University Hospitals, Atlanta, Georgia
  - Midwest Heart Foundation, Lombard, Illinois
  - Genesis Hospital Midwest Cardiovascular Research Foundation, Davenport, Iowa
  - Iowa Heart Center, West Des Moines, Iowa
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Lahey Clinic Medical Center, Burlington, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - St Joseph Mercy Hospital, Ann Arbor, Michigan
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Mercy Hospital Metropolitan Cardiology Consultants, Coon Rapids, Minnesota
  - North Mississippi Medical Center, Tupelo, Mississippi
  - Mid America Heart Institute/St. Lukes, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Bryan LGH Heart Institute, Lincoln, Nebraska
  - Morristown Memorial Hospital, Morristown, New Jersey
  - Mt Sinai Medical Center, New York, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Hospital Mid Carolinas Cardiology, Charlotte, North Carolina
  - Forsyth Medical Center, Winston-Salem, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Oklahoma Heart Hospital, Oklahoma City, Oklahoma
  - Lehigh Valley Heart Specialists, Allentown, Pennsylvania
  - Lancaster Heart & Stroke Foundation, Lancaster, Pennsylvania
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Lankenau Hospital, Wynnewood, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Spartanburg Regional, Spartanburg, South Carolina
  - Baptist Hospital, Nashville, Tennessee
  - St Thomas, Nashville, Tennessee
  - Baylor Research Institute, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Fletcher Allen Health Care, Burlington, Vermont
  - University of Virginia Health System, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - University of Wisconsin Hospital & Clinics, Madison, Wisconsin

REFERENCES:
- [Derived] Reiter MJ, Stromberg KD, Whitman TA, Adamson PB, Benditt DG, Gold MR. Influence of intracardiac pressure on spontaneous ventricular arrhythmias in patients with systolic heart failure: insights from the REDUCEhf trial. Circ Arrhythm Electrophysiol. 2013 Apr;6(2):272-8. doi: 10.1161/CIRCEP.113.000223. Epub 2013 Mar 20. PMID 23515265
- [Derived] Adamson PB, Conti JB, Smith AL, Abraham WT, Aaron MF, Aranda JM Jr, Baker J, Bourge RC, Warner-Stevenson L, Sparks B. Reducing events in patients with chronic heart failure (REDUCEhf ) study design: continuous hemodynamic monitoring with an implantable defibrillator. Clin Cardiol. 2007 Nov;30(11):567-75. doi: 10.1002/clc.20250. PMID 18000962

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began on April 28, 2006 and ended on January 14, 2011. All subjects were exited from the study on January 14, 2011. Fifty-three US clinical centers participated in the REDUCEhf study.
Pre-assignment Details: Enrolled subjects were required to have a successful implant of the Chronicle® device prior to randomization. 407 subjects had an attempted implant of the Chronicle® ICD (Implantable Cardioverter Defibrillator) (406) or Chronicle IHM (Implantable Hemodynamic Monitor) (1 subject). Of these 407 subjects, 400 were randomized.
Period: Randomized Study Period
Arm/Group | Treatment Arm | Control Arm
Started | 202 | 198
Completed | 180 | 176
Not Completed | 22 | 22
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Physician Decision | 6 | 10
Not completed — Lost to Follow-up | 4 | 0
Not completed — Death | 7 | 9
Period: Long-term Follow-up
Arm/Group | Treatment Arm | Control Arm
Started | 180 (Number entering post 12-month non-randomized long-term follow-up period) | 176 (Number entering post 12-month non-randomized long-term follow-up period)
Completed | 0 (All subjects were exited at the time of study closure) | 0 (All subjects were exited at the time of study closure)
Not Completed | 180 | 176
Not completed — Withdrawal by Subject | 9 | 9
Not completed — Physician Decision | 127 | 122
Not completed — Lost to Follow-up | 1 | 0
Not completed — Death | 14 | 11
Not completed — Study Closed | 29 | 34

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Arm | Control Arm | Total
Number analyzed (Participants) | 202 | 198 | 400
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 151 | 144 | 295
  >=65 years | 51 | 54 | 105
Age Continuous [Mean (Standard Deviation); unit: years] | 54.8 (14.7) | 54.7 (14.8) | 54.7 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 65 | 126
  Male | 141 | 133 | 274
Region of Enrollment [Number; unit: participants]
  United States | 202 | 198 | 400
NYHA (New York Heart Association) Classification [Number; unit: participants] — Class II and Class III NYHA classification
  Class II Subjects with cardiac disease resulting in slight limitation of physical activity.They are comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea, or angina.
  Class III Subjects with cardiac disease resulting in marked limitation of physical activity.They are comfortable at rest. Less than ordinary activity causes fatigue, palpitation, dyspnea, or angina.
  participants
    NYHA Class II | 107 | 90 | 197
    NYHA Class III | 95 | 108 | 203

OUTCOME MEASURES:

1. Primary Outcome: Percent of Subjects With an Attempted Implant of the Chronicle ICD System Free From System-related Chronicle ICD Complications at 6-months Post-implant.
Description: A Chronicle ICD system-related complication was defined as any system-related adverse event that occurred during the clinical investigation which is (1) treated with invasive means (including intravenous drug therapy), (2) results in death or serious injury of subject, (3) results in the explant of any Chronicle ICD component,and/or (4) causes permanent loss of significant function of the implanted system.
Time Frame: Within 6 months post-implant
Population: All 406 subjects with an attempted implant of the Chronicle ICD system.
Measure: Number (95% Confidence Interval); unit: Percentage of Chronicle ICD Subjects
Groups:
- Chronicle ICD Implanted Subjects: Analysis cohort includes all 406 subjects with an attempted implant of the Chronicle ICD system.
Arm/Group | Chronicle ICD Implanted Subjects
Number analyzed (Participants) | 406
Percentage of Chronicle ICD Subjects | 90.5 [87.7 to 93.4]
Statistical Analysis 1: Comparison: Chronicle ICD Implanted Subjects; Null hypothesis: Freedom from Chronicle system-related complications at 6-months post-implant is less than or equal to 80%. Alternative hypothesis: Freedom from Chronicle system-related complications at 6-months is greater than 80%; Test type: Superiority or Other; p < 0.001, Survival estimate at 6-months — The survival estimate at 6-months post-implant was compared to 80%. The comparison was made using the cumulative hazard [e.g. log survival estimate] for the variance; The survival estimate at 6-months post-implant was compared to 80%; 6-month survival rate = 90.5, 97.5% CI 1-sided [lower limit 87.7]

2. Primary Outcome: Percent of Subjects With an Attempted Chronicle IHM Implant Free From Chronicle IHM System-related Complications at 6-months Post-implant
Description: A Chronicle IHM system-related complication was defined as any system-related adverse event that occurred during the clinical investigation which is (1) treated with invasive means (including intravenous drug therapy), (2) results in death or serious injury of subject, (3) results in the explant of any Chronicle IHM component,and/or (4) causes permanent loss of significant function of the implanted system.
Time Frame: 6 months post implant
Population: All subjects with an attempted implant of the Chronicle IHM system were included in this analysis. At the time the study stopped, there was only one subject with an attempted Chronicle IHM implant. Thus this objective was not analyzed.
Measure: Mean (Full Range); unit: Percent of Chronicle IHM subjects
Groups:
- Chronicle IHM Implanted Subjects: Analysis cohort includes the one subject with a Chronicle IHM implant attempt
Arm/Group | Chronicle IHM Implanted Subjects
Number analyzed (Participants) | 1
Percent of Chronicle IHM subjects | 100 [100 to 100]

3. Primary Outcome: Relative Risk Reduction of All Heart Failure Related Events in the Treatment Group Compared to the Control Group
Description: The rate of HF-related events (hospitalizations >24h, hospitalizations <24h with IV therapy, ED visits with IV therapy, and urgent clinic visits with IV therapy) during the 12-month randomized follow-up period was compared between the Chronicle and Control groups.
Time Frame: 12 months post-implant
Population: All randomized subjects
Measure: Mean (95% Confidence Interval); unit: Heart failure related events per year
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 202 | 198
Heart failure related events per year | 0.48 [0.38 to 0.58] | 0.49 [0.39 to 0.59]
Statistical Analysis 1: Comparison: Treatment Arm vs Control Arm; The study was originally powered at 80% to detect a 25% risk reduction between the treatment arm and control arm with a type I error rate of 0.05. Under these assumptions 648 HF-related events from approximately 1300 subjects were required. The study stopped after 400 were randomized. Null Hypothesis: The HF-related event rate is the same between the treatment arm and control arm. Alternative Hypothesis: The HF-related event rate between the treatment arm and control arm is different; Test type: Superiority or Other; p = 0.978, Andersen-Gill — The P-value is from the Andersen-Gill model, an extension of the Cox proportional hazards model for multiple events; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.61 to 1.61] — Hazard Ratio is for the Treatment Arm relative to the Control Arm

4. Secondary Outcome: Cumulative Days in the Hospital for Heart Failure
Description: The endpoint for this objective was defined as the cumulative days in hospital for heart failure (HF) expressed as a percentage of hospital free follow-up days during the 12-month randomized period. The relatedness of the events was based on the primary reason for which the subject was originally admitted to the hospital or seen in the emergency department or at an urgent visit, not on the development of new events that occur during hospitalization.
Time Frame: 12 months post-implant
Population: All follow-up from all randomized subjects were included in this analysis.
Measure: Median (Full Range); unit: Percent days in hospital
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 202 | 198
Percent days in hospital | 0 [0 to 22] | 0 [0 to 43]
Statistical Analysis 1: Comparison: Treatment Arm vs Control Arm; Null Hypothesis: mu(Treatment) = mu(Control) Alternative Hypothesis: mu(Treatment) ne mu(Control) where mu is the percentage of hospitalized days for heart failure; Test type: Superiority or Other; p = 0.574, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Relative Risk Reduction of Cardiovascular Related Events in the Treatment Group Compared to the Control Group
Description: The rate of CV-related events (hospitalizations >24h, hospitalizations <24h with IV therapy, ED visits with IV therapy, and urgent clinic visits with IV therapy) during the 12-month randomized follow-up period was compared between the Chronicle and Control groups.
Time Frame: 12 months post-implant
Population: All randomized follow-up for all randomized subjects.
Measure: Mean (95% Confidence Interval); unit: Cardiovascular related events per year
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 202 | 198
Cardiovascular related events per year | 0.77 [0.64 to 0.89] | 0.86 [0.71 to 0.98]
Statistical Analysis 1: Comparison: Treatment Arm vs Control Arm; Null Hypothesis: The CV-related event rate is the same between the treatment arm and control arm. Alternative Hypothesis: The CV-related event rate between the treatment arm and control arm is different; Test type: Superiority or Other; p = 0.527, Andersen-Gill Model — The P-value is from the Andersen-Gill model, an extension of the Cox proportional hazards model for multiple events; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.62 to 1.28] — Hazard Ratio is for the Treatment Arm relative to the Control Arm

6. Secondary Outcome: Freedom From All Cause Death or Heart Failure Hospitalization
Description: Death from any cause or heart failure related hospitalization greater than 24 hours during the 12-month randomized period
Time Frame: 12 months post-implant
Population: All randomized subjects
Measure: Number; unit: Number of subjects meeting endpoint
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 202 | 198
Number of subjects meeting endpoint | 42 [0.73 to 0.85] | 47 [0.70 to 0.82]
Statistical Analysis 1: Comparison: Treatment Arm vs Control Arm; Null Hypothesis: Freedom from death or HF-related hospitalization is the same between the treatment arm and the control arm. Alternative Hypothesis: Freedom from death or HF-related hospitalization is different between the treatment arm and the control arm; Test type: Superiority or Other; p = 0.505, Regression, Cox; The treatment and control hazard ratio and 95% confidence interval was estimated using a univariate cox Regression Model; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.57 to 1.32] — Hazard Ratio is for the Treatment Arm relative to the Control Arm

7. Secondary Outcome: Relative Risk of All-cause Events
Description: All-cause events were defined as hospitalizations, hospitalizations <24 hours necessitating intravenous therapy, emergency department visits necessitating intravenous therapy or urgent visits necessitating intravenous therapy.
Time Frame: 12 months post-implant
Population: All randomized follow-up from all randomized subjects
Measure: Mean (95% Confidence Interval); unit: All cause event rate per year
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 202 | 198
All cause event rate per year | 1.18 [1.03 to 1.34] | 1.55 [1.36 to 1.72]
Statistical Analysis 1: Comparison: Treatment Arm vs Control Arm; Null Hypothesis: The all cause event rate is the same between the treatment arm and control arm. Alternative Hypothesis: The all cause event rate between the treatment arm and control arm is different; Test type: Superiority or Other; p = 0.088, Andersen-Gill Model; The P-value is from the Andersen-Gill model, an extension of the Cox proportional hazards model for multiple events; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.56 to 1.04] — Hazard Ratio is for the Treatment Arm relative to the Control Arm

8. Secondary Outcome: Percentage of Randomized Subjects at Each Level of the Composite Response Endpoint Between the Treatment Arm and the Control Arm.
Description: The definitions of worsened, improved, and unchanged are as follows:
  Worsened: Subject dies, is hospitalized for worsening heart failure, permanently discontinues blinded randomized assignment and has worsening heart failure at time of study discontinuation, demonstrates worsening NYHA Class at LOCF, or moderate-marked worsening of global assessment score at LOCF.
  Improved: Subject has not worsened, and demonstrates improvement in NYHA class and/or moderate-marked improvement in subject global assessment score.
  Unchanged: Subject is neither worsened nor improved.
Time Frame: 12 months post implant
Population: All randomized follow-up from all randomized subjects were included.
Measure: Number; unit: Percent of Subjects
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 202 | 198
Percent of Subjects
  Percent Subjects Improved | 51 | 51
  Percent Subjects Unchanged | 19 | 17
  Percent Subjects Worsened | 30 | 32
Statistical Analysis 1: Comparison: Treatment Arm vs Control Arm; Null Hypothesis: Distribution of composite response endpoint is the same between the treatment arm and the control arm. Alternative Hypothesis: Distribution of composite response endpoint is different between the treatment arm and the control arm; Test type: Superiority or Other; p = 0.758, Proportional odds model — P-value is from a proportional odds model comparing the distribution of composite endpoint response between the treatment arm and control arm; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.73 to 1.54] — Odds ratio represents the odds of improved score in the treatment group relative to the control group

9. Secondary Outcome: Characterize Health Resource Utilization
Description: Percentage of randomized days spent in the intensive care unit for heart failure. Reason for hospitalization was determined by the adverse event adjudication committee.
Time Frame: 12 months post implant
Population: All randomized subjects.
Measure: Mean (Full Range); unit: percentage of randomized days
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 202 | 198
percentage of randomized days | 0.1 [0 to 5.3] | 0.4 [0 to 35.1]

10. Secondary Outcome: Characterize Randomized Days Alive Out of Hospital
Description: Randomized days alive outside of the hospital was computed for each subject as the total number of randomized days minus the number of randomized days spent in the hospital for any cause.
Time Frame: 12 months post implant
Population: All randomized subjects.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 202 | 198
Days | 340 (65) | 341 (63)

11. Secondary Outcome: Characterize Subject Survival
Description: Death from any cause during the 12-month randomization period
Time Frame: 12 months post implant
Population: All randomized subjects.
Measure: Number; unit: number of deaths
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 202 | 198
number of deaths | 7 | 9
Statistical Analysis 1: Comparison: Treatment Arm vs Control Arm; Null hypothesis: Survival during the 12-month randomized follow-up period is the same between the treatment and control groups. Alternative hypothesis: Survival during the 12-month randomized period is different between the treatment and control groups; Test type: Superiority or Other; p = 0.599, Regression, Cox; The treatment to control hazard ratio and 95% confidence interval was estimated using a univariate Cox Regression Model; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.29 to 2.06] — Hazard ratio estimates the hazard of death in the treatment group relative to the control group

12. Secondary Outcome: Characterize Medication Usage
Description: The rate of change of cardiovascular medications in changes per subject month were computed and compared between treatment groups.
Time Frame: 12 months post implant
Population: All randomized subjects.
Measure: Number; unit: Medication changes per subject month
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 202 | 198
Medication changes per subject month | 1.77 | 1.49
Statistical Analysis 1: Comparison: Treatment Arm vs Control Arm; The null hypothesis is that the rate of cardiovascular medication changes is the same between the Treatment Arm and Control Arm; Test type: Superiority or Other; p = 0.145, Negative-Binomial Regression

13. Secondary Outcome: Characterize Intracardiac Pressure
Description: The average daily median estimated pulmonary arterial diastolic pressure (ePAD) was computed for each subject with at least 90 days of ePAD data available and compared between the Treatment and Control arms.
Time Frame: 12 months post implant
Population: At least 90 days of ePAD data were required for each subject during the 12-month randomized period to be included in the analysis.
Measure: Mean (Standard Deviation); unit: ePAD mm Hg
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 191 | 181
ePAD mm Hg | 22.0 (5.6) | 23.3 (6.5)
Statistical Analysis 1: Comparison: Treatment Arm vs Control Arm; Null hypothesis: Average daily median ePAD is the same between the Treatment and Control arms. Alternative hypothesis: Average daily median ePAD is the different between the Treatment and Control arms; Test type: Superiority or Other; p = 0.033, t-test, 2 sided

14. Secondary Outcome: Characterize Intracardiac Pressure Changes in Response to Subject Clinical Signs and Symptoms of Heart Failure Events
Description: The average daily median estimated pulmonary arterial diastolic pressure (ePAD) was computed for each subject with at least 90 days of ePAD data available and compared between the Control Arm subjects with and without a heart failure related event during the 12-month randomized period.
Time Frame: 12 months post implant
Population: All Control Arm subjects with at least 90 days of pressure data available during the 12-month randomized follow-up period.
Measure: Mean (Standard Deviation); unit: ePAD mm Hg
Groups:
- Heart Failure Event Free Control Subjects: Subjects randomized to the Control Arm that did not have a heart failure related event during the 12-month randomized period
- Heart Failure Event Control Subjects: Subjects randomized to the Control Arm that had a heart failure event during the 12-month randomized period
Arm/Group | Heart Failure Event Free Control Subjects | Heart Failure Event Control Subjects
Number analyzed (Participants) | 143 | 38
ePAD mm Hg | 26.3 (6.5) | 22.5 (6.3)
Statistical Analysis 1: Comparison: Heart Failure Event Free Control Subjects vs Heart Failure Event Control Subjects; Null Hypothesis: The average daily median ePAD is not different among Control Arm subjects that have and that do not have a heart failure related event during the 12-month follow-up period. Alternative Hypothesis: The average daily median ePAD is different among Control Arm subjects that have and that do not have a heart failure related event during the 12-month follow-up period; Test type: Superiority or Other; p = 0.002, t-test, 2 sided

15. Secondary Outcome: Characterize NYHA Functional Class
Description: The outcome is the change in NYHA functional class between the baseline visit and the 12-month follow-up visit. At baseline subjects were required to be NYHA functional class II or III. The outcome will show the percentage of subjects that were functional class II and III at baseline and functional class I, II, III, or IV at the 12-month visit. The percent improvement from baseline is calculated as the percentage of subjects with a lower NYHA functional class at the 12-month visit compared to their NHYA functional class at baseline.
Time Frame: baseline to 12 months post implant
Population: Subjects were required to have an NYHA functional class assessment at the baseline and 12-month follow-up visit to be included in this analysis.
Measure: Number; unit: percentage of subjects
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 177 | 173
percentage of subjects
  Percent Subjects NYHA Class II Baseline | 55 [36 to 51] | 48 [33 to 48]
  Percent Subjects NYHA Class III Baseline | 45 | 52
  Percent Subjects NYHA Class I Month 12 | 24 | 17
  Percent Subjects NYHA Class II Month 12 | 46 | 52
  Percent Subjects NYHA Class III Month 12 | 27 | 28
  Percent Subjects NYHA Class IV Month 12 | 2 | 5
  Percent Subjects Improved NYHA Class | 44 | 41
  Percent Subjects No Change in NYHA Class | 45 | 49
  Percent Subjects Worsened NYHA Class | 12 | 10
Statistical Analysis 1: Comparison: Treatment Arm vs Control Arm; Null Hypothesis: There is no difference in the change in NYHA functional class between the Treatment and Control Arms. Alternative Hypothesis: There is a difference in the change in NYHA functional class between the Treatment and Control Arms; Test type: Superiority or Other; p = 0.292, Proportional odds regression model; Odds Ratio (OR) = 1.27, 95% CI 2-sided [0.82 to 1.96] — Direction for odds ratio is the odds of improvement in the Treatment arm versus the odds of improvement in the Control arm

16. Secondary Outcome: Characterize Distance Walked in Six Minutes
Description: The outcome is the change in distance walked in 6-minutes in meters between the baseline visit and the 12-month follow-up visit. The change in distance walked was calculated within each subject as the distance walked in 6-minutes at the 12-month visit minus the distance walked in 6-minutes at the baseline visit. Positive values indicate an increase in the distance walked in 6-minutes from baseline.
Time Frame: baseline to 12 months post implant
Population: Subjects were required to complete the 6-minute hall walk test at both the baseline and 12-month visit to be included in the analysis of this objective.
Measure: Mean (Standard Deviation); unit: distance walked in 6-minutes (meters)
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 157 | 153
distance walked in 6-minutes (meters)
  Baseline visit | 313.2 (124.8) | 308.7 (133.5)
  12-month visit | 354.5 (178.8) | 347.2 (160.4)
  Change from baseline to 12-months | 41.3 (160.5) | 38.5 (154.3)
Statistical Analysis 1: Comparison: Treatment Arm vs Control Arm; Null Hypothesis: The change in 6-minute hall walk distance is not different between the Treatment and Control Arms. Alternative Hypothesis: The change in 6-minute hall walk distance is different between the Treatment and Control Arms; Test type: Superiority or Other; p = 0.996, Mixed Models Analysis

17. Secondary Outcome: Characterize Renal Function at the Baseline and 12-month Visit
Description: Change in estimated glomerular filtration rate (eGFR) from baseline to the 12-month follow-up visit. eGFR was estimated using the MDRD forumula from the National Kidney Foundation (American Journal of Kidney Diseases 39: S1-299). Change in eGFR was computed as the 12-month eGFR value minus the baseline eGFR value. Positive values indicate an increase in eGFR from baseline and negative values indicate a decrease in eGFR from baseline.
Time Frame: baseline to 12 months post implant
Population: Subjects were required to have creatinine values available at the baseline and 12-month visit to be included in the analysis of this objective.
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 175 | 173
mL/min/1.73 m^2
  Baseline eGFR | 72.4 (26.2) | 69.8 (20.4)
  12-month eGFR | 68.6 (27.7) | 69.2 (25.6)
  Change in eGFR from baseline to 12-months | -3.8 (22.0) | -0.6 (19.3)
Statistical Analysis 1: Comparison: Treatment Arm vs Control Arm; Null Hypothesis: The change from baseline to the 12-month follow-up visit in eGFR values is the same between the Treatment arm and Control arm. Alternative Hypothesis: The change from baseline to the 12-month follow-up visit in eGFR values is different between the Treatment arm and Control arm; Test type: Superiority or Other; p = 0.154, Mixed Models Analysis

18. Secondary Outcome: Characterize Intracardiac Pressure Monitoring Following Defibrillation Testing (Chronicle ICD Subjects Only)
Description: Intracardiac pressure monitoring was deemed successful following defibrillation testing if physiological pressure waveforms were present following defibrillation testing.
Time Frame: implant
Population: Of the 406 subjects with an attempted implant of the Chronicle ICD system, 366 completed defibrillation testing as part of their ICD implant procedure.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects with waveforms
Arm/Group | Chronicle ICD Implanted Subjects
Number analyzed (Participants) | 366
Percentage of subjects with waveforms | 99.7 [98.5 to 100]

19. Secondary Outcome: Characterize Defibrillation Threshold Testing Efficacy (Chronicle ICD Subjects Only)
Description: The outcome measure is the percentage of subjects implanted with the Chronicle ICD who completed defibrillation testing and had a 10 Joule safety margin
Time Frame: Implant
Population: Of the 406 subjects with an attempted implant of the Chronicle ICD system, 366 completed defibrillation testing.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Chronicle ICD Implanted Subjects
Number analyzed (Participants) | 366
percentage of subjects | 98.9 [97.2 to 99.7]

20. Secondary Outcome: Characterize Quality of Life at Baseline and 12-month Visit
Description: The outcome is the change in the Minnesota Living with Heart Failure® (MNLWHF) questionnaire response from baseline to the 12-month follow-up visit. The MNLWHF questionnaire is a 21 question questionnaire scored from zero (no impact of heart failure) to 5 (severe impact of heart failure). The composite MNLWHF score ranges from 0 (no impact of heart failure) to 105 (severe impact of heart failure). Change in MNLWHF score was computed as the 12-month minus the baseline score.
Time Frame: baseline to 12 months post implant
Population: Subjects were required to respond to the baseline and 12-month follow-up visit to be included in the analysis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 177 | 176
scores on a scale
  Baseline MNWHF score | 49.7 (26.4) | 52.7 (28.0)
  12-month MNWHF score | 34.0 (25.6) | 37.2 (25.9)
  Change in MNWHF score from baseline | -15.7 (27.3) | -15.6 (23.7)
Statistical Analysis 1: Comparison: Treatment Arm vs Control Arm; Null Hypothesis: There is no difference in the change in MNLWHF score from baseline to 12-months between the Treatment Arm and Control Arm. Alternative Hypothesis: There is a difference in the change in MNLWHF score from baseline to 12-months between the Treatment Arm and Control Arm; Test type: Superiority or Other; p = 0.583, Mixed Models Analysis; Response was change in MNLWHF score from baseline. Model adjusted for baseline MNLWHF score. Negative changes mean an improvement in MNLWHF score

21. Secondary Outcome: Characterize Arrhythmic Events
Description: The rate of spontaneous VT (ventricular tachycardia)/VF (ventricular fibrillation) episodes during the 12-month follow-up period in episodes per subject month was compared between the Treatment Arm and the Control Arm
Time Frame: 12 months post implant
Population: All 399 subjects successfully implanted with the Chronicle ICD were included in the analysis.
Measure: Number (95% Confidence Interval); unit: VT/VF episodes per subject month
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 202 | 197
VT/VF episodes per subject month | 0.54 [0.43 to 0.64] | 0.38 [0.29 to 0.47]
Statistical Analysis 1: Comparison: Treatment Arm vs Control Arm; Null Hypothesis: Rate of VT/VF episodes during the 12-month randomized period is the same between the Treatment Arm and the Control Arm. Alternative Hypothesis: Rate of VT/VF episodes during the 12-month randomized period is different between the Treatment Arm and the Control Arm; Test type: Superiority or Other; p = 0.368, Andersen-Gill Model — The P-value is from the Andersen-Gill model which adjusts for multiple VT/VF episodes per subject; Andersen-Gill model included a term for Treatment Arm. This model adjusts for multiple events per subject; Hazard Ratio (HR) = 1.48, 95% CI 2-sided [0.63 to 3.5]

ADVERSE EVENTS:
Time Frame: Time from enrollment through study closure
Description: The study collected all serious adverse events, all cardiovascular related adverse events, all adverse events related to the implanted system, and all adverse events related to the implant or system-modification procedure.
Groups:
- Enrolled, Not Randomized: 42 subjects were enrolled but exited the study prior to randomization
Arm/Group | Treatment Arm | Control Arm | Enrolled, Not Randomized
Serious Adverse Events (participants affected / at risk) | 123/202 | 136/198 | 8/42
Other Adverse Events (participants affected / at risk) | 24/202 | 25/198 | 0/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=202) | Control Arm (N=198) | Enrolled, Not Randomized (N=42)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 0 (0)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
IDIOPATHIC THROMBOCYTOPENIC PURPURA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 3 (4) | 3 (3) | 0 (0)
ANGINA PECTORIS (Cardiac disorders) | 14 (24) | 12 (16) | 0 (0)
ANGINA UNSTABLE (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 5 (5) | 10 (13) | 1 (1)
ATRIAL FLUTTER (Cardiac disorders) | 1 (3) | 2 (3) | 0 (0)
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
BRADYCARDIA (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0)
CARDIAC ARREST (Cardiac disorders) | 3 (3) | 2 (2) | 1 (1)
CARDIAC FAILURE (Cardiac disorders) | 60 (138) | 63 (166) | 4 (7)
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
CARDIOMYOPATHY (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
CORONARY ARTERY DISEASE (Cardiac disorders) | 4 (4) | 0 (0) | 0 (0)
CORONARY ARTERY STENOSIS (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
ELECTROMECHANICAL DISSOCIATION (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
LOW CARDIAC OUTPUT SYNDROME (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
MITRAL VALVE INCOMPETENCE (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 5 (6) | 0 (0) | 0 (0)
PERICARDITIS (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
SICK SINUS SYNDROME (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
SINUS ARRHYTHMIA (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
SINUS BRADYCARDIA (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
TACHYCARDIA (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
TRICUSPID VALVE INCOMPETENCE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
VENTRICULAR ARRHYTHMIA (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
VENTRICULAR FIBRILLATION (Cardiac disorders) | 5 (5) | 1 (1) | 0 (0)
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 8 (9) | 11 (12) | 0 (0)
HYPOTHYROIDISM (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
PITUITARY-DEPENDENT CUSHING'S SYNDROME (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL ADHESIONS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
COLITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
DIVERTICULAR PERFORATION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 4 (4) | 5 (5) | 0 (0)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
GINGIVAL BLEEDING (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
ILEUS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
IMPAIRED GASTRIC EMPTYING (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
PEPTIC ULCER (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
PHARYNGOESOPHAGEAL DIVERTICULUM (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
RETROPERITONEAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
UMBILICAL HERNIA, OBSTRUCTIVE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0)
CATHETER RELATED COMPLICATION (General disorders) | 0 (0) | 1 (1) | 0 (0)
CATHETER SITE HAEMATOMA (General disorders) | 1 (1) | 0 (0) | 0 (0)
DEATH (General disorders) | 2 (2) | 2 (2) | 0 (0)
HERNIA (General disorders) | 1 (1) | 0 (0) | 0 (0)
IMPLANT SITE HAEMATOMA (General disorders) | 0 (0) | 6 (6) | 0 (0)
NON-CARDIAC CHEST PAIN (General disorders) | 5 (6) | 6 (7) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 2 (2) | 0 (0)
BILE DUCT STONE (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
CHOLECYSTITIS (Hepatobiliary disorders) | 1 (1) | 3 (3) | 0 (0)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0)
PORTAL VEIN THROMBOSIS (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
TRANSPLANT REJECTION (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
ABSCESS OF EYELID (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
BACTERAEMIA (Infections and infestations) | 1 (1) | 2 (3) | 0 (0)
BACTERIAL DIARRHOEA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
BRONCHITIS (Infections and infestations) | 4 (4) | 3 (3) | 0 (0)
CELLULITIS (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
CENTRAL LINE INFECTION (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
CLOSTRIDIAL INFECTION (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
DEVICE RELATED INFECTION (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
DIVERTICULITIS (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
ENDOCARDITIS (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
GANGRENE (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 2 (2) | 4 (4) | 0 (0)
GASTROENTERITIS VIRAL (Infections and infestations) | 1 (1) | 1 (2) | 0 (0)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
IMPLANT SITE INFECTION (Infections and infestations) | 2 (2) | 3 (3) | 0 (0)
INCISION SITE INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
INFLUENZA (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
LOCALISED INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
MENINGITIS ASEPTIC (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OSTEOMYELITIS (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
PERIRECTAL ABSCESS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 8 (11) | 8 (10) | 0 (0)
PNEUMONIA STAPHYLOCOCCAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
PYELONEPHRITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
SEPSIS (Infections and infestations) | 5 (5) | 1 (1) | 1 (1)
SEPTIC SHOCK (Infections and infestations) | 3 (3) | 1 (1) | 0 (0)
TRACHEOBRONCHITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 2 (4) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
UROSEPSIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
VIRAL INFECTION (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
WOUND INFECTION (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
DEFIBRILLATION THRESHOLD INCREASED (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
DEVICE CONNECTION ISSUE (Injury, poisoning and procedural complications) | 1 (1) | 5 (5) | 0 (0)
DEVICE ELECTRICAL FINDING (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
DEVICE FAILURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
DEVICE LEAD DAMAGE (Injury, poisoning and procedural complications) | 6 (6) | 4 (4) | 1 (1)
DEVICE LEAD ISSUE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
DEVICE MALFUNCTION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
DRUG TOXICITY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
FAT EMBOLISM (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
GUN SHOT WOUND (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
INAPPROPRIATE DEVICE PROGRAMMING (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
INAPPROPRIATE DEVICE THERAPY (Injury, poisoning and procedural complications) | 4 (4) | 5 (5) | 0 (0)
INCISION SITE HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
INCISION SITE PAIN (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
LEAD DISLODGEMENT (Injury, poisoning and procedural complications) | 5 (7) | 7 (7) | 0 (0)
POST PROCEDURAL SWELLING (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
SEROMA (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
TWIDDLER'S SYNDROME (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 1 (1) | 0 (0) | 0 (0)
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 0 (0) | 3 (3) | 0 (0)
SYSTEMIC LUPUS ERYTHEMATOSUS DISEASE ACTIVITY INDEX INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
TRANSPLANT EVALUATION (Investigations) | 1 (1) | 1 (1) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 5 (5) | 4 (4) | 0 (0)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 0 (0)
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 2 (3) | 1 (1)
HYPOGLYCAEMIC SEIZURE (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 3 (6) | 0 (0) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
HYPOVOLAEMIA (Metabolism and nutrition disorders) | 6 (6) | 4 (5) | 0 (0)
OBESITY (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
COSTOCHONDRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
INTERVERTEBRAL DISC DEGENERATION (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
NEUROPATHIC ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (5) | 0 (0)
CARCINOID TUMOUR OF THE DUODENUM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
CEREBRAL HAEMANGIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
NON-SMALL CELL LUNG CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
RENAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
ALTERED MENTAL STATE LIKELY POSTICTAL (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
CAROTID ARTERY OCCLUSION (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
CAROTID ARTERY STENOSIS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 5 (5) | 1 (1) | 0 (0)
CONVULSION (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
DIZZINESS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
HEMIPARESIS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
HYPOAESTHESIA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
LACUNAR INFARCTION (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
SPINAL CORD COMPRESSION (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
SYNCOPE (Nervous system disorders) | 2 (2) | 6 (7) | 0 (0)
SYNCOPE VASOVAGAL (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
TRIGEMINAL NEURALGIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
ALCOHOL WITHDRAWAL SYNDROME (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
DEPRESSION (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0)
DEVICE PSYCHOGENIC COMPLICATION (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
MENTAL DISORDER (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
MENTAL STATUS CHANGES (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0)
SUICIDAL IDEATION (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
HAEMATURIA (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 10 (12) | 18 (18) | 3 (3)
URINARY RETENTION (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 1 (1) | 1 (1)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (2) | 0 (0)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0)
CHYLOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
PLEURISY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3) | 0 (0)
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (4) | 0 (0)
RESPIRATORY ARREST (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0)
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
SUBCUTANEOUS EMPHYSEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
AORTIC BYPASS (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
BILIARY DRAINAGE (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
CAROTID ENDARTERECTOMY (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
HEART TRANSPLANT (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0)
ILEOSTOMY CLOSURE (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
KNEE ARTHROPLASTY (Surgical and medical procedures) | 2 (2) | 3 (3) | 0 (0)
MITRAL VALVE REPLACEMENT (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
RADIOACTIVE IODINE THERAPY (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
THYROIDECTOMY (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
VERTEBROPLASTY (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
ARTERIAL STENOSIS (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
FEMORAL ARTERIAL STENOSIS (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
HYPOTENSION (Vascular disorders) | 8 (9) | 4 (4) | 1 (1)
ISCHAEMIA (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
PERIPHERAL VASCULAR DISORDER (Vascular disorders) | 3 (3) | 3 (3) | 0 (0)
THROMBOPHLEBITIS (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
THROMBOSIS (Vascular disorders) | 2 (2) | 1 (2) | 0 (0)
VENOUS OCCLUSION (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=202) | Control Arm (N=198) | Enrolled, Not Randomized (N=42)
CARDIAC FAILURE (Cardiac disorders) | 24 (45) | 25 (31) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated early after 400 of an estimated 1300 subjects required were randomized. The study was terminated due to a pressure lead integrity issue based on analysis of pressure leads from other clinical trials.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Generally, contracts allow investigators to publish study results per the protocol and publication plan. Medtronic reviews publications to determine if confidential information ("CI") is included. Any such CI is deleted before publication. Medtronic may not censor/interfere with the publication. Investigators may publish single-site publications after a decision by Medtronic that no multi-site study publication will be done or 12 months after the study is closed, whichever is earlier.